CLINICAL TRIAL: NCT02712502
Title: Open-label Comparative Safety and Efficacy Study of Levofloxacin and Amoxicillin Clavulanic Acid in Patients With Acute ,Bacterial Rhinosinusitis
Brief Title: Levofloxacin in Bacterial Rhinosinussitis
Acronym: Levolet
Status: Completed | Type: Observational
Sponsor: Dr. Reddy's Laboratories Limited (Industry)
Responsible Party: Sponsor
Other Study IDs: DRL_RUS/MD/2014/PMS/Levolet
Record Dates: First submitted 2016-03-14; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2014-11

CONDITIONS: Rhinosinusitis
MeSH Terms: conditions — Rhinosinusitis | interventions — Levofloxacin; Amoxicillin-Potassium Clavulanate Combination

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Study group (OG).: 50 patients c and acute exacerbation of chronic bacterial rhinosinusitis in the study group (OG).
  The treatment regimen in the study group.
  * Levofloxacin (Levolet) 750 mg (500 mg Levolet P + P Levolet 250 mg) 1 times a day. The course of treatment is 5 days.
  * Decongestants: xylometazoline 2 doses in each nostril two times daily - the first 5 days, then if necessary.
  Interventions: Drug: Levofloxacin
- Control group (CG).: 50 patients c and acute exacerbation of chronic rhinosinusitis in the control group (CG).
  The treatment regimen of the control group. Amoxicillin-Potassium Clavulanate Combination (875 mg of amoxicillin trihydrate, potassium clavulanate salt + 125 mg), 2 times a day. The course of treatment 10 days.
  • Decongestants: xylometazoline 2 doses in each nostril two times daily - the first 5 days, then if necessary.
  Interventions: Drug: Amoxicillin-Potassium Clavulanate Combination

INTERVENTIONS:
Drug: Levofloxacin — * Levofloxacin (Levolet) 750 mg (500 mg Levolet P + P Levolet 250 mg) 1 times a day. The course of treatment is 5 days.
  * Decongestants: xylometazoline 2 doses in each nostril two times daily - the first 5 days, then if necessary.
  Other Names: Levolet P500, Levolet P 250
  Groups: Study group (OG).
Drug: Amoxicillin-Potassium Clavulanate Combination — Amoxicillin-Potassium Clavulanate Combination (875 mg of amoxicillin trihydrate, potassium clavulanate salt + 125 mg), 2 times a day. The course of treatment 10 days.
  • Decongestants: xylometazoline 2 doses in each nostril two times daily - the first 5 days, then if necessary.
  Other Names: Amoxiclav
  Groups: Control group (CG).

SUMMARY:
Inflammatory paranasal diseases are among the most common diseases in ENT In Russia, puncture method has been conventional approach to treatment of maxillary sinusitis. However, this procedure is associated with a number of drawbacks A promising trend for the treatment of purulent sinusitis is a reasonable antibacterial therapy Fluoroquinolones, particularly levofloxacin, are highly active against pneumonocci and are more active vs. the drug products of the second generation against intracellular agents (Chlamydia spp., Mycoplasma spp., M. tuberculosis, rapidly growing atypical mycobacteria (M. avium, etc.).

Due to high activity against the agents causing bacterial upper and lower respiratory tract infections they are sometimes called "respiratory" fluoroquinolones

DETAILED DESCRIPTION:
Inflammatory diseases of paranasal sinuses occupy one of the leading positions in the overall structure of ENT-diseases.

Puncture method has been a conventional approach to the treatment of suppurative maxillary sinusitis in Russia until present. However, this relatively simple and conventional treatment method has a number of disadvantages. Fear of an unpleasant procedure is justified. Generally, single puncture does not ensure healing, and the doctor has to install drainage or of perform repeated manipulations significantly reducing quality of life during the disease period. There is also a certain risk of puncture needle penetration into adjacent areas. Sometimes direct contraindications to punctures exist (intolerance of topical anesthetics, blood clotting disorders, etc.).

The puncture itself, as an independent method, is a relieving procedure rather than a pathognomonic treatment method, especially regarding severe combined forms of sinusitis with risk of intracranial complications. Due to lacking standardized antibacterial drugs to be injected into the sinus, multiple punctures are erroneously considered to be able of eliminating the bacterial agent successfully.

One of the promising trends regarding the treatment of suppurative maxillary sinusitis is an adequate antibacterial therapy. Fluoroquinolones of last generations, levofloxacin in particular, which are highly active against pneumococci, are more effective vs. generation II drugs against intracellular agents (Chlamydia spp., Mycoplasma spp., M.tuberculosis, rapidly growing atypical mycobacteria (M.avium, etc.). At that activity towards other gram-negative bacteria is not reduced. An important property of these drugs consists in activity regarding a number of bacteria resistant to generation II fluoroquinolones. Due to high activity against the agents of upper and lower respiratory bacterial infections they are sometimes called "respiratory" fluoroquinolones.

According to a publication, Levofloxacin 500 mg q.d. for 5 days eliminated radiological signs of the disease by the end of the course in 65% subjects, while 35% showed positive changes only (М.А. Panyakina, 2012). Based on these findings, otolaryngologists have to obtain higher therapeutic efficacy levels with the same 5-day course, since this treatment term demonstrates violated compliance most frequently. One of the options is an elevation of daily dose. In particular, Rameez Shah (2013) published data concerning high efficacy of levofloxacin at a daily dose of 750 mg for 5 days.

Necessity to search ways to shorten the current course of antibiotic therapy is being under discussion at all levels. Particularly, 24th European Congress of Clinical Microbiology and Infectious Diseases performed on May 10-13, 2014 in Barcelona (ECCMID 2014) repeatedly raised question concerning revision of the current treatment standards and clinical recommendations concerning duration of antibiotic therapy and dosing regimens.

Based on the above-mentioned findings, it would be interesting to evaluate efficacy of various antibiotic schemes (respiratory fluoroquinolones or protected aminopenicillin) in hospital conditions.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form.
* Males and females aged 18-60 years old
* Hospitalized subjects with verified diagnosis of moderate/severe acute bacterial rhinosinusitis
* Readiness to comply with medical recommendations.
* Assessment of objective and subjective symptoms of the disease >= 3 points

Exclusion Criteria:

* Previous nasal surgery within the last 6 months
* Participation in other studies
* Polypous rhinosinusitis
* Concomitant therapy affecting the study results (psychotropic drugs, alpha-adrenoreceptor antagonists, antihistamine drug, antibiotics, cromones, corticosteroids) within the last month
* Need in cromones, antihistamine drugs, corticosteroids (moderate and severe allergic rhinitis)
* Severe somatic diseases in the past medical history: severe endocrine pathologies, severe cardiovascular diseases, renal and/or hepatic failure, oncology
* Subject's inability to perceive instructions for the study procedure
* Pregnancy, lactation
* Signs of a dangerous infectious disease.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: 100 Subjects with chronic bacterial rhinosinusitis were included in study. 50 subjects with acute and aggravated chronic bacterial rhinosinusitis in the main group (subjects receiving levofloxacin (Levolet® R)
  50 subjects with acute and aggravated chronic bacterial rhinosinusitis in the control group (subjects receiving levoflamoxicillin clavulanate)
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2014-09; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Reduction in mean value of Visual Analogue Scale after Levolet R therapy. TOLERABILITY of the treatment is assessed by the subjects using 10-point scale | 10 days
  Dynamics of clinical symptoms (patient assessment) disease independently evaluate patients on a 10-point system (visual analogue scale - VAS), where: 0 - no symptom, 10 points - a symptom of painful, as you can imagine.

SECONDARY OUTCOMES:
Physician's assessment: Changes in clinical symptoms using 4-point scale | 10 days
  • Dynamics of clinical symptoms (score doctor) was evaluated by a doctor of 4-point scale, where "0" - the absence of symptoms, "1" - easy to severe symptoms, "2" - moderately severe symptoms, "3" - severe symptoms.
The final evaluation of the effectiveness of treatment on | 10 days
  * "Excellent" - a significant reduction of symptoms, improvement in instrumental studies;
  * "Good" - the improvement of health, regression of symptoms, a positive trend data of laboratory and instrumental studies.
  * "satisfactory" - a slight improvement in the general condition and moderately positive dynamics of laboratory and instrumental studies.
  * "The lack of effect" - the absence of the dynamics of all symptoms, indicators of laboratory and instrumental studies, as well as when it is impossible to evaluate the effect, in the case of cessation of treatment.
  * "Deterioration" - weighting of the general condition and the negative dynamics of the indices of laboratory and instrumental studies, the need for additional treatment.
  Tolerability independently assessed patients, 10 point system, where "0" - no side effects, "10" - the inevitable need for the drug.

CONTACTS AND LOCATIONS:
Overall Officials: A Y Ovchinnikov, Principal Investigator — Head of the Department Diseases of the ear, nose and throat ,Moscow State Medical Dental University of the Ministry of Health of Russia, Otorhinolaryngology Department of Postgraduate Studies Faculty

IPD SHARING:
Plan to Share IPD: No